CLINICAL TRIAL: NCT06831721
Title: Effects of Functional Training on Vertical Jump Height, Leg Strength and Balance of the Young Volleyball Players in China.At the End of the Experiment, Functional Movement Screen, Vertical Jump, Maximum Strength of Legs and Y Balance Test Were Compared to Investigate the Effects of Non-stationary Strength Training on Youth Volleyball Players: the Non-stationary Strength Training Included the Inverted BOSU Ball Squat, Balance Capsule Single-leg Pull-up, One-legged Balance Capsule Ball Toss and Catch, and Balance Capsule Elastic Band Training
Brief Title: To Design an Experimental Intervention, 62 Youth Volleyball Players Were Divided Into an Experimental Group and a Control Group and Underwent 10 Weeks of Non-stationary Strength Training Versus Traditional Strength Training: Compared the Effects of Non-stationary Strength Training on the Athletes
Acronym: FMS、YBT、ST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, DONG KAIYUAN, Chief Researcher in UPM, Universiti Putra Malaysia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HE2024032801
Record Dates: First submitted 2025-02-11; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Unstable Strength Training; Balance Assessment
Keywords: Unstable Strength Training; balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Strength Training (Experimental): The participants' daily strength training program was interfered with by using non-stationary strength training as the intervention for the corresponding experiment.
  Interventions: Behavioral: Unstable Strength Training

INTERVENTIONS:
Behavioral: Unstable Strength Training — Sixty-two participants were divided into an experimental group and a control group. 31 participants in the experimental group were in an unstable condition, with the help of unstable equipment such as BOSU balls, balance capsules and Swiss balls. The training program was designed according to the actual situation and characteristics of the participants to meet the characteristics of the volleyball sport. The remaining 31 participants in the control group underwent a conventional strength training routine.

SUMMARY:
Purpose: Volleyball has a high influence in the world, and there are many professional volleyball players and a large number of volleyball fans in all countries. China's volleyball level ranks among the top in the world, and the Chinese women's volleyball team has won many world-class volleyball championships, but the world ranking has declined in recent years for many reasons, such as athletes' personal ability, clinical performance in the game, and injuries, etc. Functional training can effectively improve the body's functionality and reduce the risk of sports injuries. Functional training can effectively improve the body's own functionality, reduce the risk of sports injuries and thus improve the body's sports performance, while non-stationary strength training, as a kind of functional training, has little research on the effects of this training on athletes, especially youth volleyball players. In this study, inspector investigated the effects of non-stationary strength training on Functional Movement Screen (FMS), Vertical Jump Height, Leg Strength and Y Balance Test of Chinese youth volleyball players from the grassroots reserve of Chinese volleyball players.

METHODS: Sixty-four subjects participated in this experiment, 32 in the experimental group of which 18 were males and 14 were females and 32 in the control group of which 18 were males and 14 were females. The subjects were then subjected to 12 weeks of non-stationary strength training intervention in the experimental group and 12 weeks of conventional strength training in the control group, after which the pre-test, mid-test and post-test scores of FMS, Vertical Jump Height, Leg Strength and Y Balance Test were tested in the experimental and control groups. Repeated measures MANCOVA was performed using SPSS with subjects' YEAR, TALL and WEIGHT as covariates to explore changes in several dependent variables across groups and across gender. Since a female athlete in the control group was injured during the skill training in the middle of the experiment, the data of this athlete was excluded to ensure the accuracy of the data, and non-parametric tests and post hoc tests were utilized at a later stage to verify the accuracy of the repeated measures MANCOVA data.

ELIGIBILITY:
Contains Criteria:

* No congenital disorders (affecting athletic training performance)
* Meet the requirements of the FMS test
* Have a 2nd grade or higher athletic rating or two or more years of training in an athletic school
* Age 11-18 years old

Exclusion Criteria:

* Congenital heart disease
* Sports injuries that interfere with training progress prior to testing

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
The effects of non-stationary strength training on participants' Functional Movement· Screen. | From enrollment to the end of the 10-week experiment
  FMS：3 points: high-quality completion of the action. 2 points: able to complete the entire action, but compensatory action. 1 point: unable to complete the entire action or unable to maintain the starting stance.
The effects of non-stationary strength training on participants' Y Balance Test. | From enrollment to the end of the 10-week experiment
  Assuming the results are a1, b1, and c1, the composite score = (a+b+c)/(leg length * 3)* 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Liaocheng First Experimental School, Liaocheng, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided